CLINICAL TRIAL: NCT02789644
Title: A Randomized, Open-label Clinical Trial to Investigate Pharmacokinetics, Metabolomics and Biomarker in Healthy Elderly Subjects After Ursodeoxycholic Acid Administration
Brief Title: Clinical Trial to Investigate Pharmacokinetics, Metabolomics and Biomarker in Elderly After UDCA Administration
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jae Yong Chung, M.D., Ph.D, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UDCA_elderly
Record Dates: First submitted 2016-05-31; First posted 2016-06-03 (Estimated); Last update posted 2016-06-03 (Estimated); Status verified 2016-05

CONDITIONS: Aged
Keywords: Ursodeoxycholic acid; Metabolomics/biomarker; Pharmacokinetics
MeSH Terms: interventions — Ursodeoxycholic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ursodeoxycholic acid 400mg (Experimental): Day 1: Ursodeoxycholic acid 400mg qd Day 2 to 15: Ursodeoxycholic acid 200mg bid
  Interventions: Drug: Ursodeoxycholic Acid
- Ursodeoxycholic acid 800mg (Experimental): Day 1: Ursodeoxycholic acid 800mg qd Day 2 to 15: Ursodeoxycholic acid 200mg bid
  Interventions: Drug: Ursodeoxycholic Acid

INTERVENTIONS:
Drug: Ursodeoxycholic Acid — Day 1: Ursodeoxycholic acid 400mg or 800mg qd Day 2 to 15: Ursodeoxycholic acid 200mg bid
  Other Names: Ursa tab.

SUMMARY:
A clinical study to investigate pharmacokinetics, metabolomics and biomarker in healthy elderly subject after ursodeoxycholic acid administration

DETAILED DESCRIPTION:
This study has a randomized, open-label, two-treatment, one-sequence, multiple drug administration design. The purpose of this study is as follows; To investigate pharmacokinetics, metabolomics and biomarker in healthy elderly subject after ursodeoxycholic acid administration

ELIGIBILITY:
Inclusion Criteria:

* Healthy Subjects aged 70 - 84 years
* A body mass index (BMI) in the range of 18.5 kg/m2 - 29.9 kg/m2.
* Good health based on complete medical history, physical examinations, vital signs, electrocardiography (ECG), and clinical laboratory evaluations.

Exclusion Criteria:

* Subjects who have clinically significant disease of cardiovascular, respiratory, renal, endocrinological, hematological, gastrointestinal, neurological(central nervous system), psychiatric disorders or malignant tumor
* Subject judged not eligible for study participation by investigator

Ages: 70 Years to 84 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2016-05; Primary Completion 2016-07 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Area under the plasma concentration-time curve (AUC) of ursodeoxycholic acid | predose and 2, 4, 5, 7, 9, 10, 12, 24h postdose

CONTACTS AND LOCATIONS:
Overall Officials: Jae-Yong Chung, M.D., Ph.D, Principal Investigator — Department of Clinical Pharmacology and Therapeutics, Seoul National University Bundang hospital
Locations (1):
- Seoul National University Bundang Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided